CLINICAL TRIAL: NCT00183586
Title: Treatment for Adolescent Anorexia Nervosa
Brief Title: Comparing the Effectiveness of Three Types of Therapy for the Treatment of Anorexia Nervosa in Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R01MH070620 (NIH); R01MH070620 (NIH); DDTR B4-ARE
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Eating Disorders
Keywords: Treatment outcomes study; Anorexia; Anorexia nervosa
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia; Anorexia Nervosa | interventions — Family Therapy; methylcobalamin-coenzyme M methyltransferase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive family-based treatment
  Interventions: Behavioral: Family therapy (FT)
- 2 (Active Comparator): Participants will receive individual adolescent focused therapy
  Interventions: Behavioral: Individual therapy (IT)

INTERVENTIONS:
Behavioral: Family therapy (FT) — FT is a family-based treatment that will be given for a total of 24 hours over the course of 12 months.
  Other Names: FBT
  Arms: 1
Behavioral: Individual therapy (IT) — IT is an ego-oriented psychotherapy treatment that will be given for a total of 24 hours over the course of 12 months.
  Other Names: EOIT or AFT
  Arms: 2

SUMMARY:
This study will compare specific family therapy, standard family systems therapy, and standard individual psychotherapy to determine which is most effective in treating adolescent anorexia nervosa.

DETAILED DESCRIPTION:
In adolescents, anorexia nervosa severely affects physical, emotional, and social development. Despite the seriousness and prevalence of adolescent anorexia nervosa, few studies have focused on the effectiveness of various types of psychotherapy treatment. Family-based therapy may be an effective approach to treating adolescent anorexia nervosa. This study will compare specific family therapy (FT), standard family systems therapy (FS), and standard individual psychotherapy (IT) to determine which is most effective in treating adolescent anorexia nervosa. The study also aims to determine potential predictors and moderators of outcomes, as well as the cost-benefit ratio of each treatment.

Participants in this open-label study will be randomly assigned to one of three treatment groups. Group 1 will receive FT, Group 2 will receive FS, and Group 3 will receive IT. All participants will receive a total of 24 hours of their assigned therapy over a period of 12 months. Study visits will occur at baseline, immediately post-intervention, and again six months and one year post-intervention. Weight change will be assessed, as well as changes in concerns about weight and shape. The cost-benefit ratio of the treatments will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Meets Diagnostic and Statistical Manual (4th Edition) (DSM-IV) criteria for anorexia nervosa

Exclusion Criteria:

* Any psychotic illness

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 121 (Actual)
Dates: Start 2004-04; Primary Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Weight (BMI) | Measured at end-of-treatment and Months 6 and 12 post-treatment

SECONDARY OUTCOMES:
Changes in shape and weight concerns as measured with Eating Disorder Examination subscales | Measured at end-of-treatment and Months 6 and 12 post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Le Grange, PhD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States